CLINICAL TRIAL: NCT04942730
Title: Benadamustine, Fludarabine and Busulfan Conditioning in Recipients of Haploidentical Stem Cell Transplantation (FluBuBe)
Acronym: FluBuBe
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, Vice-pdirector for science RM Gorbacheva Institute, St. Petersburg State Pavlov Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06/21-n
Record Dates: First submitted 2021-06-21; First posted 2021-06-28 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Leukemia, Acute Lymphoblastic; Myeloid Leukemia, Acute; Biphenotypic Acute Leukemia; Lymphoblastic Lymphoma; Myelodysplastic Syndromes; Myeloproliferative Neoplasm
Keywords: Fludarabine; Bendamustine; Busulfan; Myeloablative Agonists; Hematopoietic Stem Cell Transplantation; Allogeneic; Antineoplastic Agents, Alkylating
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute; Myelodysplastic Syndromes; Myeloproliferative Disorders | interventions — fludarabine; Bendamustine Hydrochloride; Busulfan; Cyclophosphamide; Mycophenolic Acid; Tacrolimus; Capsules

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FluBuBe (Experimental): Days -7 through -2: Fludarabine 30 mg/m2/day iv x 6 days; Days -7 through -6: Bendamustine 130 mg/m2 iv x 2 days; Days -5 through -3: Busulfan 1 mg/kg po qid x 3 days; Days +3 through +4: Cyclophosphamide 50 mg/kg iv x 2 days; Days +5 through +35: Mycophenolate mofetil 45 mg/kg/day, maximum 3 g/day, iv or po x 30 days; Days +5 through +150: Tacrolimus 0.03 mg/kg/day with further correction by concentration
  Interventions: Drug: Fludarabine; Drug: Bendamustine Hydrochloride; Drug: Busulfan; Drug: Cyclophosphamide; Drug: Mycophenolate Mofetil; Drug: Tacrolimus 5Mg Cap

INTERVENTIONS:
Drug: Fludarabine — 30 mg/m2/day iv x 6 days, days -7 through -2 of HSCT
Drug: Bendamustine Hydrochloride — 130 mg/m2 iv x 2 days, Days -7 through -6 of HSCT
Drug: Busulfan — 1 mg/kg po qid x 3 days, Days -5 through -3
Drug: Cyclophosphamide — 50 mg/kg iv x 2 days, Days +3 through +4
Drug: Mycophenolate Mofetil — 45 mg/kg/day, maximum 3 g/day, iv or po x 30 days, Days +5 through +35
Drug: Tacrolimus 5Mg Cap — 0.03 mg/kg/day iv or po, Days +5 through +100 with with further correction by concentration. Target concentration 5-15 ng/ml.

SUMMARY:
Haploidentical hematopoietic stem cell transplantation irrespective of the conditioning and graft-versus-host disease prophylaxis is associated with high frequency of primary and secondary graft failure. Different technologies of with replete or depleted graft are associated with 10-20% of graft failures. Fludarabine and busulfan conditioning is the most commonly used approach for a variety of disease. Furthermore combination of fludarabine and bendamustine was sufficient to facilitate engraftment in patients with chronic lymphocytic leukemia and lymphomas. The aim of the study is to evaluate whether addition of bendamustine to fladarabine and busulfan conditioning reduces the risk of primary graft failure after haploidentical allograft.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have an indication for allogeneic hematopoietic stem cell transplantation with myeloablative conditioning for malignant disease
* Patients with 5-9/10 HLA-matched related donor available. The donor and recipient must be identical by the following genetic loci: HLA-A, HLA-B, HLA-Cw, HLA-DRB1, and HLA-DQB1.
* Peripheral blood stem cells or bone marrow as a graft source
* No second malignancies requiring treatment
* No severe concurrent illness

Exclusion Criteria:

* Titer of anti-HLA antibodies ≥ 5000 at the time of inclusion
* Moderate or severe cardiac dysfunction, left ventricular ejection fraction <50%
* Moderate or severe decrease in pulmonary function, FEV1 <70% or DLCO<70% of predicted
* Respiratory distress >grade I
* Severe organ dysfunction: AST or ALT >5 upper normal limits, bilirubin >1.5 upper normal limits, creatinine >2 upper normal limits
* Creatinine clearance < 60 mL/min
* Uncontrolled bacterial or fungal infection at the time of enrollment
* Requirement for vasopressor support at the time of enrollment
* Karnofsky index <30%
* Pregnancy
* Somatic or psychiatric disorder making the patient unable to sign informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
- Incidence of primary and secondary graft failure | 100 days
  Proportion of patients with primary and secondary graft failure defined by the absence of donor chimerism

SECONDARY OUTCOMES:
- Incidence of HSCT-associated adverse events (safety and toxicity) | 125 days
  Toxicity assessment is based on NCI CTC AE 5.0 grades. Veno-occlusive disease incidence and severity assessment is based on EBMT criteria 2016. Transplant-associated microangiopathy incidence assessment is based on Cho et al. criteria. All toxicity measurements will be aggregated as severity scores.
- Infectious complications, including analysis of severe bacterial, fungal and viral infections incidence | [ Time Frame: 100 days ] [ Designated as safety issue: Yes ]
  Proportion of patients, requiring systemic treatment for bacterial, viral and fungal disease
- Incidence of acute GVHD grade II-IV | 125 days
  Cumulative incidence of patients with acute GVHD II-IV grade
- Incidence of moderate and severe chronic GVHD | 365 days
  Cumulative incidence of patients with moderate and severe chronic GVHD according to NIH 2015 criteria.
- Non-relapse mortality analysis | 2 years
  Cumulative incidence of patients with mortality without hematological relapse of malignancy
- Overall survival analysis | 2 years
  Kaplan-Meier estimate of death from all causes
- Event-free survival analysis | 2 years
  Kaplan-Meier estimate of death or relapse
- Relapse rate analysis | 2 years
  Cumulative incidence of patients with relapse

CONTACTS AND LOCATIONS:
Locations (1):
- RM Gorbacheva Research Institute, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Yes
Request for sharing data with the study plan for the data will be evaluated under common conditions by Pavlov University Ethical Committee.